CLINICAL TRIAL: NCT04916431
Title: A Phase 1, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-6231, Encoding for a Human Serum Albumin - Interleukin-2 Mutein Fusion Protein (HSA-IL2m), in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-6231 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-6231-P101
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: mRNA-6231; Messenger RNA; Moderna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mRNA-6231 Dose Level 1 (Experimental): In the single dose part of the study (Sentinel and Expansion Cohorts), each participant will receive 1 dose of Dose Level 1 of mRNA-6231 by subcutaneous injection on Day 1.
  In the repeat dose part of the study (Sentinel and Expansion Cohorts), each participant will receive up to 3 doses of Dose Level 1 of mRNA-6231 once every 2 weeks.
  Interventions: Drug: mRNA-6231
- mRNA-6231 Dose Level 2 (Experimental): In the single dose part of the study (Sentinel and Expansion Cohorts), each participant will receive 1 dose of Dose Level 2 of mRNA-6231 by subcutaneous injection on Day 1.
  In the repeat dose part of the study (Sentinel and Expansion Cohorts), each participant will receive up to 3 doses of Dose Level 2 of mRNA-6231 once every 2 weeks.
  Interventions: Drug: mRNA-6231
- mRNA-6231 Dose Level 3 (Experimental): In the single dose part of the study (Sentinel and Expansion Cohorts), each participant will receive 1 dose of Dose Level 3 of mRNA-6231 by subcutaneous injection on Day 1.
  In the repeat dose part of the study (Sentinel and Expansion Cohorts), each participant will receive up to 3 doses of Dose Level 3 of mRNA-6231 once every 2 weeks.
  Interventions: Drug: mRNA-6231

INTERVENTIONS:
Drug: mRNA-6231 — Sterile frozen liquid dispersion for injection

SUMMARY:
There are 2 parts to this study: a single ascending dose (single dose of mRNA-6231) part and a multiple ascending dose (repeat doses of mRNA-6231) part. The main goal of this study is to evaluate the safety and tolerability of escalating doses of single and repeat subcutaneous (SC) administration of mRNA-6231. Dose levels of mRNA-6231 are planned to be investigated in a dose-escalation manner.

ELIGIBILITY:
Key Inclusion Criteria:

* Understand and agree to comply with the study procedures and provide written informed consent

Key Exclusion Criteria:

* Has received any investigational product (for example, study drug, biologic, device) within 30 days or 5 elimination half-lives, whichever is longer
* Pregnant or lactating women
* Men and women of childbearing potential without effective contraception during the study
* Has any lab abnormalities or clinically significant medical condition that could interfere with the interpretation of study results or limit the participant's enrollment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Up to Day 84

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of mRNA (Serum) and SM-86 (Plasma) | Predose (1 hour prior to study drug administration) to 8 hours postdose on Day 1 to Day 29
Area Under the Concentration-Time Curve (AUC) of mRNA (Serum) and SM-86 (Plasma) | Predose (1 hour prior to study drug administration) to 8 hours postdose on Day 1 to Day 29
Time to Maximum to Observed Effect (TEmax) of mRNA-6231 | Predose (1 hour prior to study drug administration) to 8 hours postdose on Day 1 to Day 29
Maximum Observed Effect (Emax) of mRNA-6231 | Predose (1 hour prior to study drug administration) to 8 hours postdose on Day 1 to Day 29
Area Under the Effect Versus Time Curve (AUEClast) of mRNA-6231 | Predose (1 hour prior to study drug administration) to 8 hours postdose on Day 1 to Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia